CLINICAL TRIAL: NCT05056272
Title: Anxiety and Sexual Malfunction in Infertile Polycystic Ovarian Syndrome Patients
Brief Title: Anxiety and Sexual Malfunction Functions in Infertile Pcos Women
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: ASMPCOSP
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS GROUP
- Non PCOS group

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common hormonal disorder in females in reproductive age associated with signs and symptoms as amenorrhea or oligomenorrhea, obesity,infertility acne and hirsutism tism that mostly Reduce self steem and having negative impact on physical and sexual quality of life , the management of signs and symptoms should result in improvement in the quality of life

ELIGIBILITY:
Inclusion Criteria:

- Age:20-40 Married infertile

Exclusion Criteria:

* any other diseases could affect quality of life

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Married infertile
Study Population: Polycystic ovary syndrome patients and infertile
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Prevellance of anxiety and sexual malfunction | 6 months
  Anticipated

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Application of female sexual function index and beck anxiety inventory for prevellance of these problems
Supporting Information: Study Protocol
Time Frame: Anticipated to be collected within 1year
Access Criteria: Married infertile women with polycystic ovary syndrome signs and symptoms

REFERENCES:
- [Result] Ehrmann DA. Polycystic ovary syndrome. N Engl J Med. 2005 Mar 24;352(12):1223-36. doi: 10.1056/NEJMra041536. No abstract available. PMID 15788499
- [Result] Hahn S, Janssen OE, Tan S, Pleger K, Mann K, Schedlowski M, Kimmig R, Benson S, Balamitsa E, Elsenbruch S. Clinical and psychological correlates of quality-of-life in polycystic ovary syndrome. Eur J Endocrinol. 2005 Dec;153(6):853-60. doi: 10.1530/eje.1.02024. PMID 16322391
- [Result] Akbari Sene A, Tahmasbi B, Keypour F, Zamanian H, Golbabaei F, Amini-Tehrani M. Differences in and Correlates of Sexual Function in Infertile Women with and without Polycystic Ovary Syndrome. Int J Fertil Steril. 2021 Jan;15(1):65-72. doi: 10.22074/ijfs.2021.6206. Epub 2021 Jan 19. PMID 33497050